CLINICAL TRIAL: NCT03778489
Title: Impact of Aerobic Exercise Training on Sympathetically Mediated Vasoconstriction and Vascular Function in Individuals With Essential Hypertension (IMPROVEH)
Brief Title: Impact of Aerobic Exercise Training on Sympathetic Vasoconstriction and Vascular Function in Essential Hypertension
Acronym: IMPROVEH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Lundbeck Foundation (Other); Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PANX-HYP
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Hypertension,Essential
Keywords: Pannexin-1 channel
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized double blinded case-control interventional study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertensive (Experimental): Men and women in age-group 35-65 years Resting blood pressure of >140/90 mmHg non or only anti-hypertensive medication
  Interventions: Other: Training
- Control (Active Comparator): Men and women in age-group 35-65 years Resting blood pressure of <140/90 mmHg no medication
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — 10 weeks of high intensity exercise training. 2-3 trainings per week of approx. 40 min.

SUMMARY:
Sympathetic nervous activity plays an important role in the development of hypertension and studies have shown that the pannexin-1 channel is involved in the signalling of the sympathetic activity to the vascular bed. The main project aim is to investigate the effects of 10 weeks of high intensity training on the effect of the sympathetic nervous activity on vascular function in individuals with essential hypertension. A secondary aim is to assess the role of essential hypertension and physical activity on vascular endothelial function,

ELIGIBILITY:
Inclusion Criteria:

* Sedentary men and women age 35 - 65 years
* Resting blood pressure >140/90 mmHg or Resting blood pressure <140/90 mmHg
* Essential hypertension
* Non or exclusively antihypertensive medication

Exclusion Criteria:

* Hypertensive condition other than essential hypertension
* Other chronical diseases
* Smoking
* Excess alcohol intake or drug abuse

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Before and after 8 weeks of training
  Changes in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Pannexin channel function assessed in vivo | Before and after 8 weeks of training
  Pannexin channel function is assessed by measurement of vascular conductance with and without channel inhibition
Pannexin channel distribution in skeletal muscle tissue | Before and after 8 weeks of training
  Pannexin channel distribution is assessed immunohistochemically in muscle samples
Sympathetic activity | Before and after 8 weeks of training
  Direct measurement of Muscle Sympathetic Nervous Activity via microneurography
Vascular function | Before and after 8 weeks of training
  Vascular conductance measured by ultrasound doppler during infusion of vasoactive substances
Mitochondrial function in endothelial cells | Before and after 8 weeks of training
  Endothelial cell mitochondrial respiration is measured by High Resolution Respirometry
Reactive oxygen species formation in in endothelial cells | Before and after 8 weeks of training
  Endothelial cell production of reactive oxygen species is measured by High Resolution Respirometry
Rheology | Before and after 8 weeks of training
  Platelet rheology. The viscoelastic measurements are based on attainment of the Gel Point (GP) from which the fractal dimension, df, is determined.
Platelet reactivity | Before and after 8 weeks of training
  Platelet reactivity is assessed by multiplate aggregometry
Maximal oxygen uptake | Before and after 8 weeks of training
  Direct Measurement of oxygen uptake during a graded test on cycle ergometer
Body Composition | Before and after 8 weeks of training
  Measured by Dual energy x-ray absorptiometry
Endothelial cell characterization | Before and after 8 weeks of training
  Assessment of protein and mRNA-levels of proteins of relevance for endothelial function
Skeletal muscle characterization | Before and after 8 weeks of training
  Assessment of protein and mRNA-levels of proteins of relevance for skeletal muscle function

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Currently awaiting instructions on this issue from the department

REFERENCES:
- [Derived] Moller S, Hansen CC, Ehlers TS, Tamariz-Ellemann A, Tolborg SAR, Kurell ME, Perez-Gomez J, Patrzalek SS, Maulitz C, Hellsten Y, Gliemann L. Exercise Training Lowers Arterial Blood Pressure Independently of Pannexin 1 in Men with Essential Hypertension. Med Sci Sports Exerc. 2022 Sep 1;54(9):1417-1427. doi: 10.1249/MSS.0000000000002936. Epub 2022 Apr 12. PMID 35420578